CLINICAL TRIAL: NCT04537845
Title: FDG PET Imaging Study of Brain Metabolic Change in Chronic Cancer Pain Patient: a Retrospective Analysis
Brief Title: Retrospective Analysis of PET Brain Imaging in Chronic Cancer Pain
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907175RINA
Record Dates: First submitted 2020-08-30; First posted 2020-09-03 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2021-08

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with cancer pain
- without cancer pain

SUMMARY:
Cancer pain deteriorated in quality of life and related with numerous psychosocial problems. Over the one third of cancer patient suffered from moderate to severe cancer pain, even under adequate pain management.

The 18F-fluoro-2-deoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) images can provide quantitative results in clinical oncology. As a functional neuroimaging, the PET evidently provided anatomical activated regions, size, and spatial extent information. In this retrospective study, we use FDG-PET to investigate changes concerning the glucose metabolism in the brain with or without cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* cancer patient

Exclusion Criteria:

* no brain metastasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patient with or without cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Find the location of brain metabolic changes, pain scale | 12 months
  This retrospective analysis only compare image and clinical record including pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Wen-ying Lin, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hosipital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin WY, Hsieh JC, Lu CC, Ono Y. Altered metabolic connectivity between the amygdala and default mode network is related to pain perception in patients with cancer. Sci Rep. 2022 Aug 18;12(1):14105. doi: 10.1038/s41598-022-18430-2. PMID 35982228